CLINICAL TRIAL: NCT01751672
Title: Integrating Substance Abuse Assessment & Intervention in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAP No. 4100055578; 09-07-05 (Other Grant/Funding Number: PA DOH)
Record Dates: First submitted 2012-12-05; First posted 2012-12-18 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Drug Use; Alcohol Use
Keywords: SBIRT; Substance Use; Screening; Brief Intervention; Primary Care
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBIRT (Active Comparator): Screening, Brief Intervention, and Referral to Treatment
  Interventions: Behavioral: SBIRT
- SBIRT+ (Experimental): Expanded Screening, Brief Intervention, and Referral to Treatment
  Interventions: Behavioral: SBIRT+

INTERVENTIONS:
Behavioral: SBIRT — Screening, Brief Intervention, and Referral to Treatment. Standard, single session SBIRT.
  Arms: SBIRT
Behavioral: SBIRT+ — Expanded Screening, Brief Intervention, and Referral to Treatment. One Standard SBIRT session, plus 2-6 additional Brief Intervention sessions as needed.
  Arms: SBIRT+

SUMMARY:
The purposes of this study are to: 1) implement a high fidelity Screening, Brief Intervention and Referral to Treatment (SBIRT) protocol with computerized screening technology into three primary care clinics in urban Philadelphia; 2) conduct a randomized controlled trial to determine if an expanded SBIRT (SBIRT+) will help patients attend more specialty substance abuse treatment sessions and reduce substance use compared to SBIRT; 3) conduct a process evaluation of SBIRT+ at the three collaborating clinics consisting of focus groups and structured interviews to assess implementation barriers and workforce attitudinal shifts; and 4) provide an excellent clinical research training environment for undergraduate and graduate students from Lincoln University.

DETAILED DESCRIPTION:
This project has several specific aims. First, investigators plan to implement a high fidelity Screening, Brief Intervention and Referral to Treatment (SBIRT) protocol with computerized screening technology into three primary care clinics in urban Philadelphia, and to train three Behavioral Health Consultants (BHCs) in an expanded brief intervention protocol (SBIRT+). Second, investigators will conduct a randomized controlled trial to address the following hypotheses: 1) patients assigned to SBIRT+ will attend more specialty substance abuse intervention and treatment sessions (excluding SBIRT+ sessions) over the 12 month follow-up than patients assigned to SBIRT; 2) patients assigned to SBIRT+ will demonstrate larger reductions in drug use by point prevalence urine samples and by reported days using over the 12-month follow-up compared to patients in SBIRT; 3) SBIRT+ will have positive net social benefits relative to SBIRT alone (i.e., will be cost-effective); 4) patients assigned to SBIRT+ will demonstrate improved medical, employment, legal, and psychiatric functioning, as well as reduced HIV risk over the 12-month follow-up compared to patients in SBIRT. Thirdly, investigators will also determine whether SBIRT and SBIRT+ are sustainable in primary care clinics as research funding for behavioral health consultants is phased out in Year 4 of the project. Investigators will also conduct a process evaluation of SBIRT+ at the three collaborating clinics consisting of focus groups and structured interviews to assess implementation barriers and workforce attitudinal shifts. This will inform methods to further disseminate SBIRT or SBIRT+, should the trial prove it is sustainable and cost-effective. Finally, investigators will provide an excellent clinical research training environment for undergraduate and graduate students from Lincoln University; this experience will balance hands-on clinical data collection and didactic training.

ELIGIBILITY:
Inclusion Criteria:

* patient is 18 years or older
* Alcohol and/or Drug screening score that indicates at least mild problem severity.

Exclusion Criteria:

* medical or psychiatric complications
* substance use is mild enough that further intervention is not warranted
* patient reports plans to leave the area within the next 12 months
* patient is unable to provide valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Session Attendance from Baseline | 0, 3, 6, 9, 12 months
  Treatment sessions attended for alcohol or drug use issues over time.

SECONDARY OUTCOMES:
Change in Urinalysis from Baseline | 0, 3, 6, 9, 12 months
  Urinalysis results for cocaine, marijuana, opiates, sedatives, and hallucinogens over time.
Change in Cost-Effectiveness from Baseline | 0, 3, 6, 9, 12 months
  Cost-effectiveness of the interventions compared to standard care over time.

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Brooks, PhD, Principal Investigator — Treatment Research Institute
Locations (3):
- United States (3):
  - Eleventh Street Family Health Services of Drexel University, Philadelphia, Pennsylvania
  - Public Health Management Corporation's Care Clinic, Philadelphia, Pennsylvania
  - Abbottsford-Falls Family Practice, Resources for Human Development, Inc., Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Chambers JE, Brooks AC, Medvin R, Metzger DS, Lauby J, Carpenedo CM, Favor KE, Kirby KC. Examining multi-session brief intervention for substance use in primary care: research methods of a randomized controlled trial. Addict Sci Clin Pract. 2016 Apr 18;11(1):8. doi: 10.1186/s13722-016-0057-6. PMID 27090097